CLINICAL TRIAL: NCT04351139
Title: Impact of the COVID-19 Pandemic on Changes in Therapeutic Strategies in Gynecological Oncology
Brief Title: Impact of the COVID-19 Pandemic in Gynecological Oncology
Acronym: COVID-GYN
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0346; 2020-A01036-33 (Other: ID-RCB)
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Gynecologic Cancer; Breast Neoplasm Female; Uterine Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms
Keywords: Gynecologic Cancer; COVID-19
MeSH Terms: conditions — Uterine Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- gynecological cancer: Patients over 18 with gynecological cancer (breast cancer, uterus, ovary, cervix, vagina or vulva cancer) and whose therapeutic management was planned during the period of COVID-19 pandemic during 2020
  Interventions: Other: modification of the planned therapeutic management
- control group: Patients over 18 with gynecological cancer (breast, uterus, ovary, cervix, vagina or vulva cancer) and whose therapeutic management was planned outside the period of COVID-19 pandemic, on the end of the year 2019
  Interventions: Other: modification of the planned therapeutic management

INTERVENTIONS:
Other: modification of the planned therapeutic management — to evaluate the changes in therapeutic management, during the COVID-19 pandemic, of patients suffering from gynecological cancers

SUMMARY:
The current infection with the Coronavirus SARS-CoV-2 (COVID-19) is an exceptional health situation which requires an adaptation of our management practices in gynecological oncology. Data from the literature suggest that infection with Coronavirus is serious in subjects with cancer with a risk of severe form 5 times higher than that of the population without cancer and a risk of death multiplied by 8. In addition, the risk of infection would be 3 times greater in case of cancer. Faced with the COVID-19 epidemic, the investigator must organize themselves to ensure continuity in the treatment of patients with gynecological cancer but also adapt our practices in the management (CPR, teleconsultation, adaptation of treatment or even postponement of treatment). The objective of the High Council of Public Health is to be able to ensure adequate oncological care avoiding any potential loss of chance concerning the care of cancer: people affected must, despite the pandemic, have care allowing the same level of curability (localized cancers) or the same life expectancy (advanced cancers). This must be done by limiting as much as possible the impact on the organization of the service, the organization of patient follow-up and the psychological impact that these possible modifications could have. The hypotheses of our study are that the exceptional health situation linked to this pandemic leads to a change in the care of patients with gynecological cancer associated with a psychological impact and increased anxiety of patients during their care. Despite the extent of the pandemic, very little existing data makes it possible to define recommendations with a sufficient level of evidence.

ELIGIBILITY:
Inclusion Criteria:

* women over 18
* gynecological cancer (breast cancer, uterus, ovary, cervix, vagina or vulva cancer)
* therapeutic management planned during quarantine
* person having expressed his non-opposition

Inclusion Criteria of control group :

* women over 18
* gynecological cancer (breast, uterus, ovary, cervix, vagina or vulva cancer)
* therapeutic management planned on the end of the year 2019
* person having expressed his non-opposition

Exclusion Criteria:

* inability to understand the information given
* person deprived of liberty,
* person under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 with gynecological cancer (non-metastatic breast cancer, uterus, ovary, cervix, vagina or vulva cancer) and whose therapeutic management was planned during the period of COVID-19 pandemic quarantine.
  Control group : Patients over 18 with gynecological cancer (breast, uterus, ovary, cervix, vagina or vulva cancer) and whose therapeutic management was planned outside the period of COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
percentage of patients with a change in the planned therapeutic management (surgery, chemotherapy, radiotherapy, hormone therapy) | Day O
  modification of the planned therapeutic management

CONTACTS AND LOCATIONS:
Overall Officials: Géry LAMBLIN, Principal Investigator — Gynaecology Department, Hôpital Femme Mère Enfant Hospices Civils de Lyon
Locations (3):
- France (3):
  - Service de Gynécologie, HFME, Hospices Civils de Lyon, Bron
  - Service de Gynécologie, Croix-Rousse, Hospices Civils de Lyon, Lyon
  - Service Gynécologie, CHLS, Hospices Civils de Lyon, Pierre-Bénite